CLINICAL TRIAL: NCT03783403
Title: A Phase 1, Open-label, Dose Finding Study of CC-95251, a Monoclonal Antibody Directed Against SIRPα, Alone and in Combination With Cetuximab or Rituximab in Subjects With Advanced Solid and Hematologic Cancers
Brief Title: A Study of CC-95251, a Monoclonal Antibody Directed Against SIRPα, in Participants With Advanced Solid and Hematologic Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-95251-ST-001; U1111-1224-8251 (Registry Identifier: WHO); NCT03816254 (obsolete NCT alias)
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neoplasms
Keywords: Antibody; CC-95251; SIRPα; Advanced Solid Cancers; Advanced Hematologic Cancers
MeSH Terms: conditions — Neoplasms | interventions — Rituximab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CC-95251 (Experimental)
  Interventions: Drug: CC-95251
- CC-95251 in combination with rituximab (Experimental)
  Interventions: Drug: CC-95251; Drug: Rituximab
- CC-95251 in combination with cetuximab (Experimental)
  Interventions: Drug: CC-95251; Drug: Cetuximab

INTERVENTIONS:
Drug: CC-95251 — Specified dose on specified days
Drug: Rituximab — Specified dose on specified days
  Arms: CC-95251 in combination with rituximab
Drug: Cetuximab — Specified dose on specified days
  Arms: CC-95251 in combination with cetuximab

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary clinical activity of CC-95251 as a single agent and in combination with cetuximab and rituximab in participants with advanced solid and hematologic cancers.

DETAILED DESCRIPTION:
This is a test.

ELIGIBILITY:
Inclusion Criteria:

* Progressed on standard anticancer therapy or for whom no other approved conventional therapy exists and have histological or cytological confirmation of advanced unresectable solid tumors, advanced unresectable colorectal cancer, or squamous cell carcinoma of the head and neck, or CD20-positive non-Hodgkin's lymphoma, or diffuse large B cell lymphoma, or follicular lymphoma
* Solid tumors must have at least one site of measurable disease as determined by RECIST v1.1
* Eastern cooperative oncology group performance status of 0 or 1

Exclusion Criteria:

* High-grade lymphomas (Burkitt's or lymphoblastic)
* Has cancer with symptomatic central nervous system (CNS) involvement
* History of class III or IV congestive heart failure (CHF) or severe non-ischemic cardiomyopathy, unstable angina, myocardial infarction, or ventricular arrhythmia within the previous 6 months

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Non-Tolerated Dose (NTD): A dose that causes unacceptable side effects | 18 months
Maximum Tolerated Dose (MTD): The highest dose that does not cause unacceptable side effects | 18 months
Dose-Limiting Toxicity (DLT): Any adverse events meeting the protocol-defined DLT criteria | 30 months

SECONDARY OUTCOMES:
Overall response rate (ORR): The percent of participants whose best response is complete response (CR) or partial response (PR) | 72 Months
Time to response (TTR): Time from the first dose to the first objective tumor response observed for participants who achieved a CR or PR | 66 Months
Duration of response (DOR): Time from the first objective tumor response observed for participants who achieved a CR or PR until the first date at progressive disease is objectively documented | 66 Months
Progression free survival (PFS): Time from the first dose to the first occurrence of disease progression or death from any cause | 66 Months
Overall survival (OS): Time from the first dose to death due to any cause | 66 Months
Pharmacokinetic - Maximum serum concentration of the drug (Cmax) | 36 Months
Pharmacokinetic - Minimum serum concentration of the drug (Cmin) | 36 Months
Pharmacokinetic - Area under the serum concentration time-curve of the drug (AUC) | 36 Months
Anti-CC-95251 antibody (ADA) assessment: determine the presence and frequency of anti-drug antibodies | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (31):
- United States (13):
  - Local Institution - 105, Birmingham, Alabama
  - Local Institution - 101, Scottsdale, Arizona
  - Local Institution - 112, Sacramento, California
  - Rocky Mountain Cancer Centers, LLP [Aurora-COAU], Aurora, Colorado
  - Local Institution - 115, St Louis, Missouri
  - Local Institution - 110, New York, New York
  - Local Institution - 109, Charlotte, North Carolina
  - Local Institution - 106, Oklahoma City, Oklahoma
  - Local Institution - 113, Portland, Oregon
  - Local Institution - 107, Pittsburgh, Pennsylvania
  - Local Institution - 102, Nashville, Tennessee
  - Local Institution - 108, Houston, Texas
  - Local Institution - 103, San Antonio, Texas
- Australia (2):
  - Local Institution - 301, Heidelberg, Victoria
  - Local Institution - 303, Melbourne, Victoria
- Canada (2):
  - Local Institution - 201, Edmonton, Alberta
  - Local Institution - 202, Toronto, Ontario
- France (6):
  - Local Institution - 402, Borddeaux Cedex
  - Local Institution - 406, Créteil
  - Local Institution - 405, Marseille
  - Local Institution - 404, Nantes
  - Local Institution - 403, Rouen
  - Local Institution - 401, Villejuif
- South Korea (4):
  - Local Institution - 604, Seoul
  - Local Institution - 603, Seoul
  - Local Institution - 602, Seoul
  - Local Institution - 601, Seoul
- Spain (3):
  - Local Institution - 504, Madrid
  - Local Institution - 502, Málaga
  - Local Institution - 501, Salamanca
- Local Institution - 802, Manchester, United Kingdom

REFERENCES:
- [Derived] Chan H, Trout CV, Mikolon D, Adams P, Guzman R, Mavrommatis K, Abbasian M, Hadjivassiliou H, Dearth L, Fox BA, Sivakumar P, Cho H, Hariharan K. Discovery and Preclinical Activity of BMS-986351, an Antibody to SIRPalpha That Enhances Macrophage-mediated Tumor Phagocytosis When Combined with Opsonizing Antibodies. Cancer Res Commun. 2024 Feb 22;4(2):505-515. doi: 10.1158/2767-9764.CRC-23-0634. PMID 38319147
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com